CLINICAL TRIAL: NCT05995938
Title: Mindfullnes-Based in Surgery Patients for Cognitive Therapy Effect
Brief Title: Mindfullnes-Based Cognitive Therapy Effect
Acronym: [Mindfullnes]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEMRA BÜLBÜLOĞLU (Other)
Responsible Party: Sponsor-Investigator, SEMRA BÜLBÜLOĞLU, Clinical Associate Professor, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022/3884
Record Dates: First submitted 2023-02-28; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Mindfullnes-Based Cognitive Therapy and Adherence to Immunosuppressive Therapy
Keywords: Liver Recipients; Transplantation; Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Experimental
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 1
  Interventions: Behavioral: Mindfullnes-Based Cognitive Therapy
- Control (No Intervention): 1

INTERVENTIONS:
Behavioral: Mindfullnes-Based Cognitive Therapy — Mindfullnes-Based Cognitive Therapy Effect on Adherence to Immunosuppressive Therapy in Liver Transplant Recipients
  Other Names: [Mindfulness]
  Arms: Experimental

SUMMARY:
Objective: In this study, the effect of mindfulness-based cognitive therapy on compliance with immunosuppressive therapy in liver transplant patients was evaluated. Method: It was conducted the study in a randomized controlled type with n=120 participation of liver transplant recipients of a transplant hospital. It was applied mindfulness-based cognitive therapy to liver recipients in the experimental group.

DETAILED DESCRIPTION:
It was used simple random sampling method in assigning liver recipients to the experimental and control groups. Discharged liver transplant patients are informed about the use of immunosuppressive drugs and the drug is prescribed. Liver transplant patients drugs.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria involved (i) being a liver transplant recipient, (ii) currently having immunosuppressive treatment, (iii) being 18 years or older (iv) having no language or communication barrier and (v) agreeing to participate in the study.

Liver transplant recipients

Exclusion Criteria:

* The exact opposite of the inclusion criteria the exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The Effect of Mindfulness-Based Cognitive after Liver Transplantation | Both groups experiment and control. It was used Mindfullnes scale and immunosuppressive terapy adherence scale. It was done measure before and after Mindfullnes-Based Cognitive Therapy.
  It will be measure Therapy on Liver Transplant Recipients' Adherence to Immunosuppressive Therapy

SECONDARY OUTCOMES:
Mindfullnes-Based Cognitive Therapy | total of six month.from 1 october 2022 to 30 Jan 2023
  le level of Mindfulness-Based Cognitive

CONTACTS AND LOCATIONS:
Locations (1):
- the Liver Transplant Hospital affiliated with Turgut Özal Medical Center of İnönü University of Malatya/Turkey., Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No